CLINICAL TRIAL: NCT06708182
Title: Social Augmentation of Self-Guided Electronic Delivery of the Life Enhancing Activities for Family Caregivers (SAGE LEAF 2): An Online Self-Guided Positive Emotion Regulation Program to Reduce Alzheimer's Dementia Caregiver Burden Delivered Through Caregiver-Serving Organizations
Brief Title: SAGE LEAF 2: An Online Program to Reduce Dementia Caregiver Burden
Acronym: SAGE LEAF 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); BrightOutcome (Industry)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor and Vice Chair for Scientific and Faculty Development, Department of Medical Social Sciences, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00222543; 2R44AG065080-03 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Caregiving Stress; Caregiver Burden
Keywords: Caregiving; Alzheimer's disease; Positive Emotion; Psychological well-being; Dementia
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Psychological Well-Being; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Positive emotion skills intervention (Experimental): Participants will go through a 6-week positive emotion skills course where 1 new skill lesson opens each week.
  Interventions: Behavioral: SAGE LEAF Positive Emotion Skills Course

INTERVENTIONS:
Behavioral: SAGE LEAF Positive Emotion Skills Course — The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access. A week will consist of 1-2 days of didactic material and 5-6 days of real-life skills practice and reporting. Participants cannot skip ahead, and can only progress to the next lesson if they have completed the current one, but they can return to old lessons or exercises if they wish to. Skills include: positive events, capitalizing, gratitude, mindfulness, positive reappraisal, personal strengths, achievable goals, self-compassion.

SUMMARY:
The goal of this clinical trial is to learn if the SAGE LEAF (Social Augmentation of self-Guided Electronic delivery of the Life Enhancing Activities for Family caregivers) online positive emotion skill-building program delivered through Caregiver Serving Organizations can help family caregivers of individuals with dementia cope with stress. The main questions it aims to answer are:

* How does SAGE LEAF affect positive emotion, caregiver burden, loneliness, and depression for family caregivers?
* What are the challenges and successes when rolling out an online program in partnership with Caregiver Serving Organizations? Participants will complete the 8-week online SAGE LEAF intervention as well as two survey assessments, one before the intervention and one after.

DETAILED DESCRIPTION:
The SAGE LEAF 2 study is a single-arm fully online implementation trial of the SAGE LEAF program delivered to family caregivers through Caregiver Serving Organizations (CSOs). The SAGE LEAF intervention is 8 weeks long and involves weekly self-guided positive emotion skill lessons, daily skill practice exercises, and daily emotion reporting, all housed on the SAGE LEAF website. The website also includes social features, such as a discussion board and profile pages, to facilitate social connection among participants. Up to n=140 family caregivers of individuals with dementia will be recruited through CSOs and the general population. To participate, caregivers must (1) identify as the primary family caregiver of a person with dementia, (2) be at least 18 years old, (3) speak and read English, and (4) have access to high-speed internet. Participants will complete survey assessments via REDCap before and after they go through the SAGE LEAF intervention. All study activities will take place online.

Individual level effectiveness will be assessed using self-reported outcomes, such as positive affect, caregiver burden, loneliness, and depression. These outcomes will be measured both pre- and post-intervention. Implementation barriers and facilitators will be assessed using follow-up qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as primary family caregiver of someone with dementia
* Speak and read English
* Has access to high speed internet and wi-fi enabled device

Exclusion Criteria:

* Care recipient lives in care facility
* Does not speak/read English
* Does not have access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden measured using the Zarit Burden Interview. | Baseline and 8 weeks
  Assesses perceived burden in caregivers by assessing subjective feelings of the impact of caregiving on emotional and physical health, financial strain, and social functioning. Scale values range from "Never" to "Nearly Always" with higher scores reflect greater burden.
Positive Aspects of Caregiving measured using the Positive Aspects of Caregiving scale | Baseline and 8 weeks
  11-item scale that identifies positive consequences of caregiving, such as feeling more useful, feeling appreciated, and strengthening relationships with others. Values range from "Disagree a lot" to "Agree a lot." Higher scores indicate greater identification of the positives of being a caregiver.
Positive Affect measured using the PROMIS Bank v1.0 Positive Affect | Baseline and 8 weeks
  Computer adaptive test (CAT) that assess momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement, over the past 7 days, using a scale of not at all to very much, where higher scores indicate higher levels of positive emotion.
Caregiver self-efficacy/mastery measured using the Caregiving Mastery subscale of the Caregiving Appraisal Measure | Baseline and 8 weeks
  12-item Caregiving Mastery subscale of the Caregiving Appraisal Measure. Values range from "Disagree a lot" to "Agree a lot" and "Never" to "Nearly Always" with higher scores indicating higher feelings of caregiving mastery.
Anxiety measured by PROMIS Bank v1.0 Anxiety | Baseline and 8 weeks
  Computer adaptive test (CAT) that assesses level of anxiety by having participants rate items focused on depressive symptoms over the past 7 days, using scale from Never to Always, where higher scores indicate higher levels of anxiety.
Depression measured by PROMIS Bank v1.0 Depression | Baseline and 8 weeks
  Computer adaptive test (CAT) that assesses depressive mood by having participants rate items focused on depressive symptoms over the past 7 days, using scale from Never to Always, where higher scores indicate higher levels of depression.
Social isolation measured by PROMIS Bank v2.0 Social Isolation | Baseline and 8 weeks
  Computer adaptive test (CAT) that assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Values range from Never to Always, and higher scores indicate higher degree of social isolation.
Self-efficacy measured by PROMIS Bank v1.0 General Self-Efficacy | Baseline and 8 weeks
  Computer adaptive test (CAT) that assesses ones confidence in their ability to succeed in specific situations or complete a task. Values range from "I am not at all confident" to "I am very confident", where higher scores indicate higher confidence.
Life satisfaction measured by PROMIS Bank v1.0 General Life Satisfaction | Baseline and 8 weeks
  Computer adaptive test (CAT) assesses one's cognitive evaluation of life experiences and whether one likes his/her life or not. Values range from "Strongly disagree" to "Strongly agree" with higher scores indicating higher degrees of satisfaction with one's life.
Perceived stress measured by Cohen's Perceived Stress Scale | Baseline and 8 weeks
  Ten item scale that measure the degree to which situations in one's life are appraised as stressful. Respondents are asked to indicate how often they felt or thought a certain way during the last month on a scale of 0 (Never) to 4 (Very Often), with higher scores indicating higher levels of perceived stress.
Perceived social support measured by the Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline and 8 weeks
  12-item measure of perceived adequacy of social support from three sources: family, friends, & significant other; using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree), where higher scores indicate higher perceptions of social support.
Meaning and Purpose measured using PROMIS Bank v1.0 Meaning and Purpose | Baseline and 8 weeks
  Computer adaptive test (CAT) assesses the degree to which one feels life has purpose and there are good reasons for living, including hopefulness, optimism, goal-directedness, and feelings that one's life is worthy. Scale values range from "Strongly disagree" to "Strongly agree" on items 1-3, and "Not at all" to "Very much" on items 4-8, with higher values associated with a higher sense of meaning and purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States